CLINICAL TRIAL: NCT07318441
Title: Determinants of Functional Capacity in Patients With Fibromyalgia
Brief Title: Functional Capacity Determinants in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Betül Taşpınar, Prof. Dr., Izmir Democracy University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FMS-35
Record Dates: First submitted 2025-12-23; First posted 2026-01-06 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Fibromyalgia; Fatigue
Keywords: fibromyalgia; functional capacity; fatigue
MeSH Terms: conditions — Fibromyalgia; Fatigue

STUDY DESIGN:
Intervention Model Description: Individuals diagnosed with fibromyalgia according to the American College of Rheumatology criteria
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fibromyalgia Group (Other): Patients diagnosed with fibromyalgia who attend the Physical Medicine and Rehabilitation Outpatient Clinic will undergo comprehensive assessments of functional capacity, pain, fatigue, mobility, muscle strength, posture, psychosocial factors, physical activity level, circadian rhythm, and sleep quality. No intervention will be applied.
  Interventions: Other: Assessment Only

INTERVENTIONS:
Other: Assessment Only — No therapeutic intervention will be applied. Participants will undergo standardized clinical, functional, and self-reported assessments, including functional capacity tests, pain and fatigue evaluation, mobility and muscle strength assessments, posture analysis, psychosocial questionnaires, physical activity level, circadian rhythm, and sleep quality evaluation

SUMMARY:
Fibromyalgia is a chronic pain disorder characterized by widespread pain and multiple systemic symptoms that negatively affect functional capacity. Although common symptoms and clinical features of fibromyalgia have been well described, the factors influencing functional capacity remain unclear. Therefore, this study aims to identify the determinants of functional capacity in patients with fibromyalgia.

DETAILED DESCRIPTION:
Fibromyalgia is a chronic pain disorder characterized by widespread pain, fatigue, sleep disturbances, cognitive problems, and mood disorders, affecting 5% of the population, predominantly women. This condition lacks objective diagnostic markers and relies on subjective symptoms and tender points for diagnosis. The etiology of fibromyalgia, which involves biological, genetic, and environmental factors, remains unclear, making diagnosis difficult due to symptom variability and comorbidities. Pathophysiological mechanisms are not fully understood, leading to difficulties in diagnosis and treatment. Historically, fibromyalgia has evolved from terms such as 'neurasthenia' to 'fibrositis', and understanding has shifted from muscle inflammation to central nervous system dysfunction. The American College of Rheumatology criteria play a crucial role in diagnosing fibromyalgia, helping to reduce patient anxiety and unnecessary testing. In the literature, pain, fatigue, sleep problems, and trigger point sensitivity are among the symptoms frequently seen in fibromyalgia patients. Studies conducted on these symptoms indicate that patients particularly experience anxiety, depression, decreased functional capacity, decreased functional mobility, postural abnormalities, decreased respiratory and peripheral muscle strength, decreased physical activity, and difficulties in daily living activities.

Although surveys conducted with fibromyalgia patients have identified symptoms, no studies have been found that examine the factors affecting functional capacity. Therefore, the aim of this study is to determine the factors affecting functional capacity in patients with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with fibromyalgia according to the American College of Rheumatology criteria
* Be 18 years of age or older
* Be a volunteer
* Be able to read and write

Exclusion Criteria:

* Having a condition that prevents communication,
* Having undergone surgery within the last 6 months
* Being an elite athlete
* Having an active infection
* Having a neurological or orthopedic problem that prevents movement
* Being a cancer patient

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (for Pain and Fatigue) | baseline
  Pain intensity and fatigue intensity will be assessed using the visual analog scale (VAS). It is frequently preferred because it is an easy and understandable scale. Participants are asked to mark the appropriate place on a 10 cm horizontal line, where the beginning indicates no pain and the end indicates unbearable pain. The same scale will be used to assess fatigue intensity. The beginning of the line indicates no fatigue, and the end indicates extreme fatigue. To measure the intensity, the distance from the beginning of the line to the point marked by the participant will be measured with a ruler and recorded
6-Minute Walk Test | baseline
  The 6-minute walk test is a reliable test for fibromyalgia patients and has been used as an indicator of cardiorespiratory fitness in patients with fibromyalgia. It is frequently used in the assessment of functional capacity. It is simple, practical, and inexpensive. It does not require special equipment or advanced training and is well tolerated by patients. The patient is asked to walk as fast as they can without running in a corridor of at least 30 meters. The distance covered in 6 minutes is measured.
Timed Up and Go Test | baseline
  It is a reliable test frequently used to assess agility, dynamic balance, and functional mobility in individuals with fibromyalgia. The Timed Up and Go test was developed by Podsiadlo and Richardson (1991). Participants will begin the test by sitting in a chair with back support. They will stand up from the chair, walk to a mark 3 meters away, and return to sit down, at which point the time will be recorded .
30-second sit-to-stand test | baseline
  Used to measure lower body muscle strength. Participants begin the test by sitting on a chair with their arms crossed at chest level and their hands on their shoulders. From this sitting position, they must stand up until their knees are fully extended and then sit back down until their backs touch the back of the chair. The number of repetitions within 30 seconds is recorded. It is a reliable test for individuals with fibromyalgia
Hand Grip Strength | baseline
  Grip strength is considered an indicator of upper extremity muscle strength. Measurements will be recorded by testing the dominant and non-dominant hand three times using the JAMAR hand dynamometer. This device is a widely used and highly reliable grip strength measurement tool. The test will be performed in a sitting position, with the upper arm parallel to the body, the elbow flexed at 90 degrees, and the forearm and hand in a neutral position.
Assessment of Tender Points | baseline
  In our study, an algometer device will be used to assess tender points. The algometer device is a reliable device that can be used to assess tender points. Eighteen tender points will be assessed according to the American College of Rheumatology criteria for the classification of fibromyalgia. They will be marked with a pen before use. The tender points to be marked are: occipital, lower cervical, trapezius, supraspinatus, second rib, lateral epicondyle, gluteal, greater trochanter, and knees. Pain assessment will be performed by applying a vertical pressure of approximately 1 kg/s to the tender points with the algometer, and the person will be asked to report when the pressure becomes painful. A high algometer score indicates low pain
New York Posture Assessment | baseline
  The New York Posture Assessment is a valid and reliable assessment used in posture evaluation. Posture is assessed from the lateral and posterior views. It includes a series of three-digit drawings for each of the 13 body alignment sections. These are scored as 5 (correct posture), 3 (mild deviation), or 1 (significant deviation). The highest score is 65, and the lowest is 13. A score ≥45 is "excellent," 40-44 is "good," 30-39 is "moderate," 20-29 is "poor," and ≤19 is "very poor"
Revised Fibromyalgia Impact Questionnaire | baseline
  A study by Ediz and colleagues demonstrated that the Turkish version of the Revised Fibromyalgia Impact Questionnaire is a reliable and valid tool. It is a self-reported questionnaire that measures functional capacity and disease severity in patients with fibromyalgia. It is an easy and short questionnaire. It consists of 3 sections with 21 questions on function, overall impact, and symptoms. It concerns experiences in the last 7 days and is scored using an 11-point numerical rating scale. The total score for the function domain (range 0 to 90, divided by 3), the global impact domain score (range 0 to 20), and the symptoms domain score (range 0 to 100, divided by 2)
Multidimensional Fatigue Inventory | baseline
  Smets et al. developed the Multidimensional Fatigue Inventory-20 (MFI-20), which consists of five fatigue subscales: general fatigue, physical fatigue, mental fatigue, decreased motivation, and decreased activity. It has been used in various descriptive and experimental studies of many different diseases, including fibromyalgia. Özilhan et al.'s study demonstrated that the Turkish oncology version of the MFI-20 is a valid and reliable measure of fatigue in cancer patients, while Başoğlu et al.'s study demonstrated that it is a valid and reliable measure of fatigue in patients with multidimensional FM. When completing the scale, individuals are asked to select the degree closest to themselves, ranging from "no, not true" to "yes, very true." It consists of 20 questions. A high score indicates severe fatigue.
Fibromyalgia Participation Questionnaire | baseline
  This is a scale that evaluates patients' social participation, daily life, and work life over the past four weeks. The questionnaire consists of 27 items. The first 16 items relate to daily life, and the following 6 items focus on the patients' social lives. Item 23 asks patients whether they are currently employed, and they can answer with "yes" or "no". Patients who answer "yes" are then asked about the level of difficulty they experience in their work life on five separate items. Patients are allowed to rate these levels on a scale of 1 to 5. The total score is calculated as the sum of the first 22 items for patients who are not employed, and as the sum of all 27 items for patients who are employed. The minimum score for those who are not employed is 22, and the maximum score is 110; for those who are employed, the minimum score is 27, and the maximum score is 135. A higher score indicates a more severe impairment (restriction).
Pain Catastrophizing Scale | baseline
  This is a self-administered questionnaire used to assess the patient's feelings and thoughts about pain. It was developed by Sullivan and colleagues in 1995. It is a reliable and valid Turkish-language questionnaire that assesses specific variables such as severe pain, disability, and emotional distress following trauma or tissue damage. It consists of the subscales "helplessness" (inability to cope effectively with pain), 'magnification' (dissatisfaction caused by excessive focus on the negative consequences of pain), and "rumination" (inability to stop thinking about pain). It consists of 13 items and is scored on a scale of 0 to 4. It is a 52-point scale.
Kinesiophobia Assessment | baseline
  Participants in our study will be assessed for kinesiophobia, or fear of movement/re-injury, using the Tampa Kinesiophobia Scale, whose test-retest reliability in Turkish has been demonstrated by Tunca Yılmaz and colleagues. The scale was first developed in 1991 but was not published. It was published by Vlaeyen and colleagues in 1995. The scale covers work-related activities, injury/re-injury, and fear-avoidance. It consists of 17 questions. It is scored as follows: Strongly disagree 1, Disagree 2, Agree 3, Strongly agree 4. It is scored between 17 and 68. The higher the score, the higher the fear of movement.
Hospital Anxiety and Depression Scale | baseline
  It consists of 14 questions in total, 7 of which assess anxiety, 7 assess depression, and the odd-numbered questions assess anxiety symptoms while the even-numbered questions assess depression symptoms. Each question is scored between 0 and 3. Higher scores indicate higher levels of anxiety and depression.
Circadian Rhythm Assessment | baseline
  The Morningness-Eveningness Questionnaire was developed by Horne and Ostberg in 1976 to behaviorally assess individuals' circadian rhythms and interpersonal biological rhythm variations [39]. It is the most commonly used measure for assessing chronotype preference.It consists of 19 self-assessment items, and scores are calculated according to five chronotype categories. A high score indicates a strong morning preference.
International Physical Activity Questionnaire Short Form (IPAQ) | baseline
  It is a commonly used measure for assessing physical activity. In our study, the 7-item International Physical Activity Questionnaire Short Form will be used.The number of days and duration of vigorous physical activity, moderate physical activity, and walking activities lasting at least 10 minutes or longer in the past 7 days are assessed. The number of days and minutes are calculated by multiplying each activity's MET value. Vigorous physical activities are calculated as 8 MET, moderate physical activities as 4 MET, and walking as 3.3 MET. Time spent sitting is not included in the scoring. All are added together for the overall physical activity score. A weekly MET value below 600 is considered inactive, 601-3,000 is moderately active, and above 3,000 is active.
Pittsburgh Sleep Quality Index | baseline
  This is a questionnaire consisting of 24 questions that assesses individuals' sleep quality and sleep disorders.The first 19 questions are answered by the individual themselves, while the last 5 questions are to be answered by their spouse or roommate. The last 5 questions are not included when calculating the total score. A high score indicates poor sleep quality. The first 19 questions assess a wide range of factors to estimate sleep duration, sleep onset latency, and the frequency and severity of sleep-related problems. It consists of a total of 7 subheadings: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disorders, use of sleep medications, and daytime dysfunction. Each subheading is scored from 0 to 3 and has its own calculation method. The total score ranges from 0 to 21. A score of 5 or above indicates poor sleep quality .

CONTACTS AND LOCATIONS:
Overall Officials: Beyzanur Beğenen Şavlı, Msc.Pt., Principal Investigator — Izmir Democracy University; Betül Taspinar, Prof.Dr., Principal Investigator — Izmir Democracy University; Ferruh Taspinar, Prof.Dr., Principal Investigator — Izmir Democracy University
Locations (1):
- Betül TAŞPINAR, Konak, İ̇zmi̇r, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No